CLINICAL TRIAL: NCT04124965
Title: A Randomized, Open-Label Extension Study to Investigate the Long-Term Safety, Tolerability, and Efficacy of Rozanolixizumab in Adult Patients With Generalized Myasthenia Gravis
Brief Title: A Study to Investigate the Long-term Safety, Tolerability, and Efficacy of Rozanolixizumab in Adult Patients With Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG0004; 2019-000969-21 (EudraCT Number)
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Generalized Myasthenia Gravis
Keywords: UCB7665; generalized myasthenia gravis; rozanolixizumab; gMG
MeSH Terms: conditions — Myasthenia Gravis | interventions — rozanolixizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rozanolixizumab dosage regimen 1 (Experimental): Study participants randomized to dosage regimen 1 will receive assigned dosage of rozanolixizumab at pre-specified time points during the Treatment Period. The dose regimen may be switched based on investigator discretion.
  Interventions: Drug: Rozanolixizumab
- Rozanolixizumab dosage regimen 2 (Experimental): Study participants randomized to dosage regimen 2 will receive assigned dosage of rozanolixizumab at pre-specified time points during the Treatment Period. The dose regimen may be switched based on investigator discretion.
  Interventions: Drug: Rozanolixizumab

INTERVENTIONS:
Drug: Rozanolixizumab — Rozanolixizumab will be administered by subcutaneous infusion in dosage regimen 1 or 2.
  Other Names: UCB7665

SUMMARY:
The purpose of the MycarinGstudy is to evaluate the long-term safety, tolerability and long-term efficacy of rozanolixizumab in study participants with generalized myasthenia gravis (MG).

ELIGIBILITY:
Inclusion Criteria:

* Participant was eligible for MG0003 [NCT03971422] or MGC003 at the time of enrollment into either study and the participant either completed the observation Period of MG0003 or MGC003 or required rescue therapy during the Observation Period of the lead-in studies
* Body weight ≥35 kg at Visit 1
* Study participants may be male or female

Exclusion Criteria:

* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, if applicable, chest X-rays (posterior anterior and lateral), and TB testing by a positive (not indeterminate) QuantiFERON®-TB Gold Plus
* Participant has received a live vaccination within 8 weeks prior to the Baseline visit; or intends to have a live vaccination during the course of the study or within 8 weeks following the final dose of study medication
* Study participant has experienced hypersensitivity reaction after exposure to other anti-neonatal Fc receptor (FcRn) drugs - Study participant with severe (defined as Grade 3 on the myasthenia gravis-activates of daily living (MG-ADL) scale) weakness affecting oropharyngeal or respiratory muscles, or who has myasthenic crisis or impending crisis
* Participant has any laboratory abnormality that, in the opinion of the Investigator, is clinically significant, has not resolved at randomization, and could jeopardize or compromise the study participant's ability to participate in this study
* Study participant met any mandatory withdrawal or mandatory study drug discontinuation criteria MG0003 [NCT03971422] or MGC003, or discontinued study medication in either study, with the exception of discontinuation due to a need for rescue treatment
* Study participant is not considered capable of adhering to the protocol visit schedule, or medication intake according to the judgment of the Investigator
* Study participant has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or had suicidal ideation since the last visit in MG0003 as indicated by a positive response (Yes) to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 22733 (UCB)
Locations (43):
- United States (10):
  - Mg0004 50081, Phoenix, Arizona
  - Mg0004 50072, Los Angeles, California
  - Mg0004 50088, Washington D.C., District of Columbia
  - Mg0004 50120, Miami, Florida
  - Mg0004 50073, Tampa, Florida
  - Mg0004 50114, Indianapolis, Indiana
  - Mg0004 50121, Lexington, Kentucky
  - Mg0004 50077, New York, New York
  - Mg0004 50090, Winston-Salem, North Carolina
  - Mg0004 50096, Philadelphia, Pennsylvania
- Canada (3):
  - Mg0004 50066, Montreal
  - Mg0004 50070, Québec
  - Mg0004 50069, Toronto
- Czechia (2):
  - Mg0004 40125, Ostrava-Poruba
  - Mg0004 40124, Prague
- Mg0004 40128, Aalborg, Denmark
- France (4):
  - Mg0004 40129, Bordeaux
  - Mg0004 40132, Nice
  - Mg0004 40133, Paris
  - Mg0004 40131, Strasbourg
- Germany (3):
  - Mg0004 40140, Göttingen
  - Mg0004 40078, Leipzig
  - Mg0004 40177, Münster
- Italy (4):
  - Mg0004 40144, Milan
  - Mg0004 40146, Pavia
  - Mg0004 40148, Roma
  - Mg0004 40150, Roma
- Japan (5):
  - Mg0004 20078, Hanamaki Shi
  - Mg0004 20079, Hiroshima
  - Mg0004 20077, Miyagi
  - Mg0004 20076, Shinjuku-Ku
  - Mg0004 20032, Suita
- Poland (3):
  - Mg0004 40155, Gdansk
  - Mg0004 40154, Lodz
  - Mg0004 40151, Lublin
- Russia (4):
  - Mg0004 20027, Moscow
  - Mg0004 20001, Saint Petersburg
  - Mg0004 20028, Saint Petersburg
  - Mg0004 20055, Saint Petersburg
- Spain (2):
  - Mg0004 40159, Barcelona
  - Mg0004 40157, L'Hospitalet de Llobregat
- Taiwan (2):
  - Mg0004 20080, Taichung
  - Mg0004 20081, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this study may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Derived] Bril V, Druzdz A, Grosskreutz J, Habib AA, Kaminski HJ, Mantegazza R, Sacconi S, Utsugisawa K, Vu T, Boehnlein M, Gayfieva M, Greve B, Woltering F, Vissing J; MG0004 study investigators. Safety and efficacy of chronic weekly rozanolixizumab in generalized myasthenia gravis: the randomized open-label extension MG0004 study. J Neurol. 2025 Mar 19;272(4):275. doi: 10.1007/s00415-025-12958-9. PMID 40105996
- [Derived] Bril V, Druzdz A, Grosskreutz J, Habib AA, Mantegazza R, Sacconi S, Utsugisawa K, Vissing J, Vu T, Boehnlein M, Bozorg A, Gayfieva M, Greve B, Woltering F, Kaminski HJ; MG0003 study team. Safety and efficacy of rozanolixizumab in patients with generalised myasthenia gravis (MycarinG): a randomised, double-blind, placebo-controlled, adaptive phase 3 study. Lancet Neurol. 2023 May;22(5):383-394. doi: 10.1016/S1474-4422(23)00077-7. PMID 37059507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in Oct 2019 and concluded in Sep 2021.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Groups:
- Rozanolixizumab ~7 mg/kg: Participants received rozanolixizumab equivalent to approximately 7 milligrams/kilogram (mg/kg), subcutaneously on a weekly basis over a 52-week Treatment Period. After 52-week Treatment Period, participants were followed up for 8 weeks (up to Week 60).
- Rozanolixizumab ~10 mg/kg: Participants received rozanolixizumab equivalent to approximately 10 mg/kg, subcutaneously on a weekly basis over a 52-week Treatment Period. After 52-week Treatment Period, participants were followed up for 8 weeks (up to Week 60).
Period: Overall Study
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Started | 35 | 36
Safety Set (Received at least 1 dose of investigational medicinal product) | 35 | 35
Completed | 5 | 3
Not Completed | 30 | 33
Not completed — Adverse event, non-fatal | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Rolled Over To MG0007 Study | 25 | 28
Not completed — Pregnancy | 1 | 0
Not completed — Sponsor and participant decision | 0 | 1
Not completed — Personal surgery | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) which consisted of all study participants who were randomized, using the treatment assigned instead of the actual treatment received.
Groups:
- Rozanolixizumab ~7 mg/kg: Participants received rozanolixizumab equivalent to approximately 7 mg/kg, subcutaneously on a weekly basis over a 52-week Treatment Period. After 52-week Treatment Period, participants were followed up for 8 weeks (up to Week 60).
- Total: Total of all reporting groups
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 26 | 55
  >=65 years | 6 | 10 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (14.2) | 53.7 (17.2) | 52.2 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 16 | 17 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 4 | 8
  Black | 2 | 3 | 5
  White | 17 | 19 | 36
  Missing | 12 | 10 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 19 | 25 | 44
  Missing | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an AE starting on or after the time of first administration of investigational medicinal product (IMP) or any unresolved event already present before the first administration of IMP that worsened in intensity following exposure to IMP, up to 8 weeks after the last dose of IMP in study participants who discontinued the study or IMP.
Time Frame: From Baseline until End of Study (up to Week 60)
Population: The Safety Set (SS) consisted of all randomized study participants who received at least 1 dose of IMP in this study. This endpoint was planned to be analyzed using the SS by most recent dose received i.e. the most recent dose received at or before the AE onset. Participants who switched doses were counted in both rozanolixizumab (RLZ) doses.
Measure: Number; unit: percentage of participants
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 50 | 42
percentage of participants | 76.0 | 78.6

2. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Permanent Withdrawal of Study Medication
Description: A TEAE is defined as an AE starting on or after the time of first administration of IMP or any unresolved event already present before the first administration of IMP that worsened in intensity following exposure to IMP, up to 8 weeks after the last dose of IMP in study participants who discontinued the study or IMP.
Time Frame: From Baseline until End of Study (up to Week 60)
Population: The Safety Set consisted of all randomized study participants who received at least 1 dose of IMP in this study. This endpoint was planned to be analyzed using the SS by most recent dose received i.e. the most recent dose received at or before the AE onset. Participants who switched doses were counted in both rozanolixizumab doses.
Measure: Number; unit: percentage of participants
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 50 | 42
percentage of participants | 6.0 | 0

3. Secondary Outcome: Change From Baseline in Myasthenia Gravis-Activities of Daily Living (MG-ADL) Total Score at Each Scheduled Assessment During Treatment and Observation Periods
Description: The Myasthenia Gravis Activities of Daily Living (MG-ADL) is an 8-item patient-reported outcome (PRO) instrument developed on the basis of the Quantitative Myasthenia Gravis (QMG). The MG-ADL targeted symptoms and disability across ocular, bulbar, respiratory, and axial symptoms. The total MG-ADL score was obtained by summing the responses to each individual item (8 items; Grades: 0, 1, 2, 3), where 0 represents no symptoms or impaired performance and 3 represents the most severe symptoms or impaired performance. The total score ranges from 0 to 24, with a higher score indicating more disability. A positive change indicates worsening and a negative change indicates improvement.
Time Frame: Baseline, Weeks 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 52 and 60
Population: The Safety Set consisted of all randomized study participants who received at least 1 dose of IMP in this study. Here, number analyzed signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 35 | 35
units on a scale
  Week 5: number analyzed (Participants) | 34 | 34
  Week 5 | -2.7 (3.3) | -3.2 (3.8)
  Week 7: number analyzed (Participants) | 35 | 32
  Week 7 | -2.7 (3.8) | -3.7 (3.4)
  Week 9: number analyzed (Participants) | 29 | 31
  Week 9 | -2.8 (3.4) | -3.4 (3.7)
  Week 13: number analyzed (Participants) | 30 | 30
  Week 13 | -3.1 (3.4) | -3.9 (4.0)
  Week 17: number analyzed (Participants) | 25 | 29
  Week 17 | -2.8 (3.3) | -4.0 (3.9)
  Week 21: number analyzed (Participants) | 20 | 24
  Week 21 | -3.0 (3.4) | -4.1 (4.3)
  Week 25: number analyzed (Participants) | 18 | 17
  Week 25 | -2.7 (3.0) | -3.7 (4.7)
  Week 29: number analyzed (Participants) | 13 | 14
  Week 29 | -2.8 (2.1) | -3.6 (4.3)
  Week 33: number analyzed (Participants) | 10 | 12
  Week 33 | -3.0 (2.8) | -3.5 (4.5)
  Week 37: number analyzed (Participants) | 7 | 10
  Week 37 | -3.9 (2.5) | -3.6 (3.6)
  Week 41: number analyzed (Participants) | 6 | 6
  Week 41 | -2.8 (2.1) | -1.8 (1.0)
  Week 45: number analyzed (Participants) | 4 | 7
  Week 45 | -3.8 (2.4) | -2.1 (1.1)
  Week 49: number analyzed (Participants) | 5 | 6
  Week 49 | -2.4 (1.1) | -0.5 (3.7)
  Week 52: number analyzed (Participants) | 5 | 3
  Week 52 | -2.6 (1.3) | -2.0 (NA) — NA signifies that as pre-specified in the Statistical Analysis Plan, Standard Deviation was only calculated if there were a minimum of 4 participants.
  Week 60: number analyzed (Participants) | 7 | 7
  Week 60 | -0.3 (2.1) | -1.3 (3.9)

4. Secondary Outcome: Change From Baseline in Myasthenia Gravis-Composite (MG-C) Total Score at Each Scheduled Assessment During Treatment and Observation Periods
Description: MG-C scale is a validated assessment and scale tests 10 items with individual items being weighted differently. The items included ptosis/upward gaze (range: 0 [>45 second] - 3 [Immediate]), double vision on lateral gaze (range: 0 [>45 second] - 4 [Immediate]), eye closure (range: 0 [Normal] - 2 [severe weakness]), talking (range: 0 [Normal] - 6 [difficult to understand speech]), chewing (range: 0 [Normal] - 6 [gastric tube]), swallowing (range: 0 [Normal] - 6 [gastric tube]), breathing (range: 0 [Normal] - 9 [ventilator dependence]), neck flexion (range: 0 [Normal] - 4 [severe weakness]), shoulder abduction (range: 0 [Normal] - 5 [severe weakness]) and hip flexion (range: 0 [Normal] - 5 [severe weakness]), lower scores= lower disease activity. Total MG-C score was obtained by summing responses to each individual item and score ranges from 0 to 50, with lower scores indicating lower disease activity. A positive change indicates worsening and a negative change indicates improvement.
Time Frame: Baseline, Weeks 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 52 and 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 35 | 35
units on a scale
  Week 5: number analyzed (Participants) | 34 | 35
  Week 5 | -4.7 (5.5) | -5.5 (7.3)
  Week 7: number analyzed (Participants) | 35 | 33
  Week 7 | -5.0 (5.7) | -7.1 (7.4)
  Week 9: number analyzed (Participants) | 29 | 30
  Week 9 | -5.0 (5.3) | -6.0 (7.4)
  Week 13: number analyzed (Participants) | 30 | 30
  Week 13 | -4.8 (5.5) | -7.0 (7.8)
  Week 17: number analyzed (Participants) | 25 | 29
  Week 17 | -4.4 (5.7) | -5.5 (8.6)
  Week 21: number analyzed (Participants) | 20 | 24
  Week 21 | -5.3 (6.9) | -7.3 (8.1)
  Week 25: number analyzed (Participants) | 18 | 17
  Week 25 | -6.1 (5.8) | -8.8 (7.7)
  Week 29: number analyzed (Participants) | 13 | 14
  Week 29 | -5.1 (5.5) | -9.1 (9.2)
  Week 33: number analyzed (Participants) | 9 | 12
  Week 33 | -4.6 (5.1) | -8.4 (8.6)
  Week 37: number analyzed (Participants) | 7 | 10
  Week 37 | -6.3 (6.8) | -8.6 (6.9)
  Week 41: number analyzed (Participants) | 6 | 6
  Week 41 | -6.0 (7.1) | -6.5 (5.8)
  Week 45: number analyzed (Participants) | 4 | 7
  Week 45 | -4.0 (6.2) | -5.3 (4.9)
  Week 49: number analyzed (Participants) | 5 | 6
  Week 49 | -1.4 (3.8) | -0.8 (9.2)
  Week 52: number analyzed (Participants) | 5 | 2
  Week 52 | -3.8 (3.1) | NA (NA) — NA signifies that as pre-specified in the Statistical Analysis Plan, mean was only calculated if there were a minimum of 3 participants and standard deviation was only calculated if there were a minimum of 4 participants.
  Week 60: number analyzed (Participants) | 7 | 7
  Week 60 | 1.7 (3.7) | -2.3 (8.5)

5. Secondary Outcome: Change From Baseline in Quantitative Myasthenia Gravis (QMG) Total Score at Each Scheduled Assessment During Treatment and Observation Periods
Description: The QMG is a validated assessment and the scale tested 13 items, including ocular and facial involvement, swallowing, speech, limb strength, and forced vital capacity. The total QMG score was obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3) and the score ranges from 0 to 39, with lower scores indicating lower disease activity. A positive change indicates worsening and a negative change indicates improvement.
Time Frame: Baseline, Weeks 5, 7, 9, 13, 17, 21, 25, 29, 33, 37, 41, 45, 49, 52 and 60
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 35 | 35
units on a scale
  Week 5: number analyzed (Participants) | 34 | 34
  Week 5 | -2.9 (4.7) | -4.5 (4.4)
  Week 7: number analyzed (Participants) | 35 | 32
  Week 7 | -3.3 (4.4) | -5.2 (4.3)
  Week 9: number analyzed (Participants) | 28 | 30
  Week 9 | -3.3 (3.8) | -4.7 (4.3)
  Week 13: number analyzed (Participants) | 30 | 29
  Week 13 | -2.6 (4.2) | -5.5 (4.4)
  Week 17: number analyzed (Participants) | 25 | 28
  Week 17 | -3.1 (4.9) | -4.2 (4.4)
  Week 21: number analyzed (Participants) | 20 | 23
  Week 21 | -4.0 (4.7) | -5.1 (4.9)
  Week 25: number analyzed (Participants) | 18 | 16
  Week 25 | -5.1 (4.6) | -5.7 (5.5)
  Week 29: number analyzed (Participants) | 13 | 13
  Week 29 | -5.4 (3.6) | -5.5 (6.3)
  Week 33: number analyzed (Participants) | 10 | 11
  Week 33 | -4.9 (4.8) | -6.2 (5.7)
  Week 37: number analyzed (Participants) | 7 | 9
  Week 37 | -5.3 (3.9) | -6.8 (5.9)
  Week 41: number analyzed (Participants) | 6 | 5
  Week 41 | -5.7 (4.3) | -4.0 (3.1)
  Week 45: number analyzed (Participants) | 4 | 6
  Week 45 | -5.3 (2.8) | -4.0 (3.5)
  Week 49: number analyzed (Participants) | 5 | 5
  Week 49 | -3.8 (0.8) | -1.8 (1.8)
  Week 52: number analyzed (Participants) | 5 | 2
  Week 52 | -4.6 (2.9) | NA (NA) — NA signifies that as pre-specified in the Statistical Analysis Plan, mean was only calculated if there were a minimum of 3 participants and standard deviation was only calculated if there were a minimum of 4 participants.
  Week 60: number analyzed (Participants) | 7 | 6
  Week 60 | -0.9 (2.4) | -1.8 (5.1)

6. Secondary Outcome: Percentage of Participants Using Rescue Medication (Intravenous Infusion of Immunoglobulin G (IVIg) or Plasma Exchange (PEX))
Description: Rescue therapy consisted of IVIg or PEX. Study participants who experienced disease worsening (eg, an increase of 2 points on the MG-ADL or 3 points on the QMG scale between 2 consecutive visits) may be considered for rescue therapy at the discretion of the Investigator.
Time Frame: From Baseline until End of Study (up to Week 60)
Population: The Safety Set consisted of all randomized study participants who received at least 1 dose of IMP in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
Number analyzed (Participants) | 35 | 35
percentage of participants | 11.4 | 0

ADVERSE EVENTS:
Time Frame: From Baseline until End of Study (up to Week 60)
Description: TEAEs are reported in the safety section. TEAEs were planned to be analyzed using the SS by most recent dose received i.e. the most recent dose received at or before the AE onset. Participants who switched doses were counted in both RLZ doses.
Arm/Group | Rozanolixizumab ~7 mg/kg | Rozanolixizumab ~10 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/42
Serious Adverse Events (participants affected / at risk) | 7/50 | 2/42
Other Adverse Events (participants affected / at risk) | 27/50 | 25/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rozanolixizumab ~7 mg/kg (N=50) | Rozanolixizumab ~10 mg/kg (N=42)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Biopsy kidney abnormal (Investigations) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 3 (4) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rozanolixizumab ~7 mg/kg (N=50) | Rozanolixizumab ~10 mg/kg (N=42)
Diarrhoea (Gastrointestinal disorders) | 6 (11) | 7 (10)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (8)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4)
Pyrexia (General disorders) | 4 (5) | 3 (4)
Hypogammaglobulinaemia (Immune system disorders) | 2 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2)
Blood immunoglobulin G decreased (Investigations) | 6 (12) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 15 (55) | 12 (40)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT04124965/Prot_001.pdf
  • Statistical Analysis Plan (2021-09-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT04124965/SAP_002.pdf